CLINICAL TRIAL: NCT06807723
Title: Further Delineation of the De Santo Shinawi Syndrome Phenotype Using a Series of Individuals Carrying a Pathogenic Variant of the WAC Gene
Acronym: 2024-CF366
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-CF366
Record Dates: First submitted 2024-11-14; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-11

CONDITIONS: WAC; DeSanto-Shinawi Syndrome; DESSH; WAC SYNDROME; OMIM#616708; ORPHA:466943
Keywords: Further delineation of the De Santo Shinawi Syndrome; Serie of patients with DESSH; Better characterization of DeSanto-Shinawi Syndrome; Series of individuals with pathogenic WAC variant; WAC; DeSanto; DeSanto-Shinawi; De Santo Shinawi; DESSH; OMIM 616708; OMIM#616708; ORPHA:466943; ORPHA 466943

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Serie of patients with a molecular diagnosis of DeSanto-Shinawi Syndrome

SUMMARY:
The aim of this retrospective, multicenter study would be to extend the phenotypic spectrum of DeSanto Shinawi Syndrome and improve the knowledge of its evolution. To this end, the investigators would like to issue a call for international collaboration in order to create a series of new genetically diagnosed patients, not yet described in previous publications, and with a larger number of individuals evaluated in a single study. One of the aims would be to establish a set of standardized clinical and paraclinical examinations to be carried out at diagnosis and for follow-up of affected patients. This would enable patients, their families and the caregivers involved to better anticipate future management.

DETAILED DESCRIPTION:
Main objective :

Update clinical and paraclinical knowledge of DeSanto-Shinawi syndrome.

Secondary objectives:

* Inventory the clinical signs of the syndrome described to date and look for recurrence between patients.
* Select a set of standardized clinical and paraclinical examinations for diagnosis.
* Establish appropriate management and follow-up.
* To compare the phenotype of patients with DESSH due to a pathogenic point variation in the WAC gene and those with a microdeletion involving the WAC gene.

Main inclusion criteria:

Children and adults of any age. Molecular diagnosis of a pathogenic variant involving the WAC gene (SNV, CNV, SV).

Main non-inclusion criteria:

Patients with a molecular diagnosis of another VP (SNV) of a gene responsible for a neurodevelopmental disorder.

Patient having already participated in a DESSH study with published data. No patient data available.

Primary endpoint:

The data collected will enable the investigators to meet the objective, namely to expand clinical and paraclinical knowledge of DeSanto-Shinawi syndrome.

Main secondary endpoints: NA (descriptive study) Statistics: NA (descriptive study)

ELIGIBILITY:
Inclusion Criteria:

* Children and adults of any age.
* Molecular diagnosis of a pathogenic (or likely pathogenic) variant involving the WAC gene (SNV, CNV, SV).

Exclusion Criteria:

* Patients with a molecular diagnosis of another VP (SNV) of a gene responsible for a neurodevelopmental disorder.
* Patient having already participated in a DESSH study with published data.
* No patient data available.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of any age with a molecular and clinical diagnosis of DeSanto-Shinawi Syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Clinical knowledge | Through study completion, an average of 2 years
  Morphologic description with photos (optional) at a specified date (front and side of the face, hands-feet : plant and palm) using HPO terms
Clinical knowledge | Through study completion, an average of 2 years
  Overall clinical examination and interrogatory at the last medical consultation (neurologic, cardiologic, gastroenterologic, pulmonary, urinary, global development, etc.) : data collected using a redcap form.
Clinical knowledge | Through study completion, an average of 2 years
  Height, weight and head circumferance at birth and at last visit
Paraclinical knowledge | Through study completion, an average of 2 years
  Any psychometric scale performed during lifetime : Language delay, Motor delay, ADHD, IQ, ASD
Paraclinical knowledge | Through study completion, an average of 2 years
  Any exams performed during lifetime : EEG, neuroMRI, abdominal echography, cardiac echography

SECONDARY OUTCOMES:
Recurrence of clinical signs | Through study completion, an average of 2 years
  Inventory the clinical signs of the syndrome described to date and mesure concordance or not
Standardized examinations | Through study completion, an average of 2 years
  Using concordance of signs, mesure the clinical and paraclinical necessary at diagnosis
Management & Follow-up | Through study completion, an average of 2 years
  Using concordance of signs at different ages, establish appropriate management and follow-up.
Genotype phenotype correlation | Through study completion, an average of 2 years
  Compare the phenotype of DESSH patients with pathogenic point variation in the WAC gene and those with microdeletion involving the WAC gene

CONTACTS AND LOCATIONS:
Overall Officials: Florian CHERIK, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Clermont-Ferrand University Hospital, Clermont-Ferrand, Auvergne, France

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.

REFERENCES:
- See also: Patients with DeSanto-Shinawi syndrome: Further extension of phenotype from Italy; Pasquali et al. — https://pubmed.ncbi.nlm.nih.gov/36420948/